CLINICAL TRIAL: NCT03447119
Title: Living Well With a Disability Curriculum Adaptation Evaluation Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Southern University (Other)
Responsible Party: Principal Investigator, Gavin Colquitt, Associate Professor, Georgia Southern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H18234
Record Dates: First submitted 2018-01-31; First posted 2018-02-27 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Health Education; Community Health Services; Health Services for Persons With Disabilities; Developmental Disabilities
MeSH Terms: conditions — Health Education; Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Living Well with a Disability (Experimental): The parents will work together with the project directors to deliver the adapted curriculum to participating families. With bi-weekly meetings for 10 weeks between parent facilitators and family participants in the home or another desired location. The project directors have already participated in the facilitator training and will serve as mentors to newly trained facilitators. At the end of the online training session, the parent facilitators will be equipped to successfully implement the Living Well curriculum.
  Interventions: Behavioral: Living Well with a Disability

INTERVENTIONS:
Behavioral: Living Well with a Disability — Implementation of an adapted health promotion program.

SUMMARY:
The purpose of this proposal is to implement a joint project with Georgia Southern University and the Effingham County Navigator Team to improve the quality of life of families with a child with a disability in southeast Georgia. The final outcome of this project will be a new curriculum, Living Well Together, which builds on a previous implementation of the Living Well with a Disability curriculum in Bulloch County.

DETAILED DESCRIPTION:
First, parent facilitators will be recruited and matched with their peers. Parent facilitators will be members of the Effingham County Navigator Team with a child with a disability. The peer matching resembles the community lay health worker model. The community lay health worker model will reduce the amount of time needed to meet face to face with families. To begin adapting the facilitator training and curriculum, the program directors will work with representatives from the University of Montana Rural Institute on Disabilities to review and update training materials. A representative from the Rural Institute on Disabilities will deliver an online intensive facilitator training. The facilitator training is approximately 15 hours long. The training includes three major components: peer training, facilitator training, and Master "Train the Trainer" training. The project directors will work with the Effingham County Navigator Team to recruit parents. The Navigator Team will recruit five parents as parent facilitators. The parents will work together with the project directors to deliver the adapted curriculum to participating families. With bi-weekly meetings for 10 weeks between parent facilitators and family participants in the home or another desired location. The project directors have already participated in the facilitator training and will serve as mentors to newly trained facilitators. At the end of the online training session, the parent facilitators will be equipped to successfully implement the Living Well curriculum. The project directors will schedule a working meeting before and after the facilitator training to discuss curriculum changes with the Rural Institute on Disabilities representative. Changes in readability are anticipated since the target audience includes adolescents. Curriculum delivery methods will need tailoring to match a family-based approach including activities to be completed at the home at the family and individual levels for parents, siblings, and children. Both GSU faculty and the Navigator team will lead monthly summary meetings to review the adapted content. These meetings will take place at a convenient location in the community as determined by the Navigator team. Pre and post focus groups will take place before and after these monthly meetings at a convenient locale in the community.

ELIGIBILITY:
Inclusion Criteria

Families of with a child (3-50) with any developmental disability

Exclusion Criteria

Family and child are unable to follow directions and participate in curriculum activities.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-03-24 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Global Health | 12 months
  Patient Reported Outcomes Measurement Information System Parent Proxy scale v 1.0
  Global Health
  * Patient Reported Outcome Measurement Information System (PROMIS) Pediatric Global Health (PROMIS PGH-7) measures general health, quality of life, physical health, mental health, feeling sad, social health (fun with friends), and parents listening to ideas.
  * Each item is measured on a likert scale from 1 (never) to 5 (always). There is one item for each subscale listed above. A range for each subscale would be 1-5. Typically, results are reported as a whole so the range would be 7 to 35.
  * For each subscale and the scale as a whole the higher the score, the better the global health.
  * Subscales are summed to compute the total score.

SECONDARY OUTCOMES:
Family Relationships | 12 months
  Patient Reported Outcomes Measurement Information System Parent Proxy scale v. 1.0
  Family Relationships
  * The Family Relationships subscale measures the importance and strength of the family unit perceived by the child in the past four weeks.
  * Each item is measured on a Likert scale from 1 (never) to 4 (always). There are four items in this subscale. The reports are reported as a whole so the range is 4 to 16.
  * The higher the score, the stronger the family relationships.
  * Items are summed for the total score.
Life Satisfaction | 12 months
  Patient Reported Outcomes Measurement Information System Parent Proxy scale v 1.0 Life Satisfaction
  * The Life Satisfaction subscale measures quality of life in the past four weeks.
  * Each item is measured on a Likert scale from 1 (not at all) to 5 (very much). There are eight items in this scale. The range for the whole subscale is 8-40.
  * The higher the score, the better quality of life.
  * Each item is summed for the total score.
Physical Activity | 12 months
  Patient Reported Outcomes Measurement Information System Parent Proxy scale v 1.0 Physical Activity
  * The Physical Activity subscale reports frequency and intensity of exercise of the child in the past week.
  * Each item is measured on a Likert scale from 1 (no days) to 5 (6-7 days). There are eight items in this subscale. The total range is 8 (no exercise) to 40 (exercising regularly).
  * The higher the score, the more physically active the individual is.
  * The items are summed together for the score.
Psychological Stress Experiences | 12 months
  Patient Reported Outcomes Measurement Information System Parent Proxy scale v 1.0 Psychological Stress Experiences
Peer Relationships | 12 months
  Patient Reported Outcomes Measurement Information System Parent Proxy scale v 1.0 Peer Relationships
  * The Peer Relationships subscale measures the child's social activity in the last 7 days.
  * Each item is measured on a Likert scale from 1 (never) to 5 (almost always). There are 7 items in the scale. The range is 7 (doesn't interact with friends) to 35 (very socially active).
  * The higher the score the better the relationships.
  * The items are summed together for a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Colquitt, EdD, Principal Investigator — Georgia Southern University
Locations (1):
- B and B Care Services, Springfield, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT03447119/Prot_SAP_000.pdf